CLINICAL TRIAL: NCT07122583
Title: Study to Collect Post-Market Data on Non-Invasive Subcutaneous Fat Reduction in the Submental, Inner Thigh and Back/Bra Areas With the CoolSculpting Elite System
Brief Title: A Study to Assess Non-Invasive Subcutaneous Fat Reduction in the Submental, Inner Thigh and Back/Bra Areas With the CoolSculpting Elite System
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-970; ZA24-002 (Other: AbbVie)
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Non-Surgical Fat Reduction
Keywords: Non-Surgical Fat Reduction; CoolSculpting Elite System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cohort A: Submental (Other): Participants will receive applications of the CoolSculpting Elite System in the submental body area.
  Interventions: Device: CoolSculpting Elite System
- Cohort B: Inner Thigh (Other): Participants will receive applications of the CoolSculpting Elite System in the inner thigh (bilateral) body area.
  Interventions: Device: CoolSculpting Elite System
- Cohort C: Back/Bra (Other): Participants will receive applications of the CoolSculpting Elite System in the back/bra (bilateral) body area.
  Interventions: Device: CoolSculpting Elite System

INTERVENTIONS:
Device: CoolSculpting Elite System — CoolSculpting Elite Applicator

SUMMARY:
The primary objective of this protocol is the continued collection of data specific to the submental, inner thigh and back/bra body areas with CoolSculpting Elite. The study aims to collect post-market safety data while allowing for the collection of standardized photos and satisfaction questionnaires after treatment with commercial treatment parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participant has clearly visible fat on the submental, bilateral inner thigh or bilateral back/bra areas, which in the investigator's opinion, is appropriate for treatment with CoolSculpting Elite.
* Participant has not had weight change exceeding 5% of body weight in the preceding month.

Exclusion Criteria:

* Participant has had a recent surgical procedure in the area of intended treatment within the previous 6 months.
* Participant has had previous surgical or invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Participant has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the previous 12 months.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Device and/or Procedure-Related Adverse Events (AEs) | Up to Approximately 6 Months
  Frequency of device and procedure-related AEs including serious device-related adverse events (SADEs), will be analyzed per cohort.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Pacific Clinical Innovations, Vista, California, United States

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-970